CLINICAL TRIAL: NCT04088812
Title: Interventional Trial to Evaluate a Meat Derivative Product and a Satiating Compound on Satiety in a Group of Healthy Overweight Subjects
Brief Title: Meat Derivative and Satiating Compound Effect on Satiety
Acronym: SACIMEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Creaciones Aromáticas Industriales, S.A. (CARINSA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HULP 5389
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Overweight
Keywords: Satiety; Meat derivative; Fiber; Visual Analogue Scale; Parallel
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo meat derivative + Placebo satiating compound (Placebo Comparator): 60 g Placebo meat derivative 25 g Placebo satiating compound
  Interventions: Other: Placebo meat derivative + Placebo satiating compound; Other: Placebo meat derivative + Satiating compound; Other: Experimental meat derivative + Placebo satiating control
- Placebo meat derivative + Satiating compound (Experimental): 60 g Placebo meat derivative 25 g Satiating compound
  Interventions: Other: Placebo meat derivative + Placebo satiating compound; Other: Placebo meat derivative + Satiating compound; Other: Experimental meat derivative + Placebo satiating control
- Experimental meat derivative + Placebo satiating control (Experimental): 60 g Experimental meat derivative 25 g Placebo satiating compound
  Interventions: Other: Placebo meat derivative + Placebo satiating compound; Other: Placebo meat derivative + Satiating compound; Other: Experimental meat derivative + Placebo satiating control

INTERVENTIONS:
Other: Placebo meat derivative + Placebo satiating compound — Subjects will consume 60 g of meat derivative placebo in a brunch type meal with 25 g of the satiating compound placebo diluted in water
Other: Placebo meat derivative + Satiating compound — Subjects will consume 60 g of meat derivative placebo in a brunch type meal with 25 g of the satiating compound diluted in water
Other: Experimental meat derivative + Placebo satiating control — Subjects will consume 60 g of the experimental meat derivative in a brunch type meal with 25 g of satiating compound placebo diluted in water

SUMMARY:
The purpose of this study is to evaluate the satiating effects of a meat derivative and a satiating compound on overweight subjects (BMI ≥25 and <30 kg / m2).

DETAILED DESCRIPTION:
A randomized, parallel, controlled and double-blind pilot study with 3 study arms is being performed to evaluate the satiating properties of a meat derivate and a satiating compound in a group of healthy overweight subjects.

The investigators included 20 participants between 18 and 65 years (BMI ≥25 and <30 kg / m2). All volunteers will be randomized into 3 study groups, and participants will receive the 2 study products during the 3 experimental phases.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 65 years old.
* Body Mass Index (BMI) ≥25 and <30 kg/m2.
* Adequate cultural level and understanding for the clinical trial.
* Subjects willing to consume all food present in the brunch type meal.
* Signed informed consent.

Exclusion Criteria:

* Subjects with BMI ≥30 or <25 kg /m2. Subjects with a vegetarian diet or with a great fiber consumption (> 30 g/day)
* Subjects diagnosed with Diabetes Mellitus.
* Subjects with dyslipidemia on pharmacological treatment.
* Subjects with hypertension on pharmacological treatment.
* Subjects with hyper/hypothyroidism.
* Subjects with established diagnosis of eating disorder.
* Smokers or those subjects with high alcohol consumption (> 2-3 servings/day in men and> 1 serving/day in women (1 serving = 1 glass of wine or 1 bottle of beer).
* Subjects under pharmacological treatment (except oral contraceptives).
* Subjects with large weight fluctuations of more than 4 kg or who have undergone in six months a weight loss diet.
* Subjects with gastrointestinal diseases that affect the digestion or absorption of nutrients.
* Subjects with severe chronic diseases (hepatic, kidney, …)
* Subjects with intense physical activity.
* Subjects with food allergies to meals included in breakfast, study product or lunch or that reject their consumption.
* Subjects with a diagnosis of celiac disease or a gluten intolerance.
* Subjects who consume regularly oral supplements (i.e. omega-3)
* Pregnant or breastfeeding women.
* Women with menstrual irregularities (absence of menstrual cycle at least 2 months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 10 men and 10 women
Enrollment: 19 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Satiety Hunger Assessment | 0 min to 240 min
  Visual Analogue Scale (VAS). 100 mm horizontal line anchored at each end with the extremes of the subjective feeling to be quantified. Subjects are instructed to rate the sensation being experienced according to how they define the line.
  e.g., "not at all hungry" (0mm) and "as hungry as I have ever felt" (100mm). Multiple measures are taken at repeated time intervals described below.

SECONDARY OUTCOMES:
Change from Baseline Blood Hormonal Satiety Markers | 0 min to 240 min
  Glucagon-like peptide-1 (GLP-1), Peptide tyrosine-tyrosine (YY), Ghrelin, Leptin, Gastric Inhibitory Peptide (GIP), Peptide C
Amount of food consumed in a "food ad libitum" | 240 min
  240 min After eating the study product
Total amount of food consumed in 24h | 24 hours
  24h Food Record Method
Change from Baseline Glucose Metabolism Parameters | 0 min to 240 min
  Concentration of Glucose
Anthropometric Parameters | 24 hours
  Weight and height will be combined to report BMI in kg/m2
Adverse Effects | 24 hours
  Number of participants with gastrointestinal symptoms (Nausea, Diarrhea, Bloating and other disorders)

CONTACTS AND LOCATIONS:
Overall Officials: Bricia López Plaza, PhD, Principal Investigator — La Paz University Hospital
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain